CLINICAL TRIAL: NCT07281469
Title: Comparison of the Functional Outcomes of Closed Reduction and Plaster of Paris Application Versus Closed Reduction With K-Wire Fixation and Plaster of Paris Application in the Management of Colles' Fracture.
Brief Title: Comparison of Functional Outcomes of Closed Reduction With Cast Versus Closed Reduction With K-Wire Fixation in Colles' Fracture
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khawaja Muhammad Safdar Medical College (Other)
Responsible Party: Principal Investigator, Suqlain Ali, Dr Suqlain Ali post graduate resident, Khawaja Muhammad Safdar Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMSafdarMC
Record Dates: First submitted 2025-11-18; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Colles' Fracture
MeSH Terms: conditions — Colles' Fracture

STUDY DESIGN:
Intervention Model Description: There are two groups in the study each group contains 30patients ,group A apply plaster of Paris for colles fracture and group B patients treated with k wires and plaster of Paris
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Closed Reduction and Plaster of Paris Cast Application (Active Comparator): Closed reduction followed by Plaster of Paris cast application
  Interventions: Procedure: Closed reduction and fracture manipulation and plaster of Paris application in group A
- Closed Reduction with Percutaneous K-Wire Fixation and Plaster of Paris Cast Application (Active Comparator): Closed Reduction With K-Wire Fixation and POP Cast Closed reduction followed by percutaneous K-wire fixation and Plaster of Paris cast application
  Interventions: Procedure: closed reduction and Percutaneous K-wire fixation and plaster of application is applied in group B

INTERVENTIONS:
Procedure: Closed reduction and fracture manipulation and plaster of Paris application in group A — Closed reduction and manipulation of fracture and application of plaster of Paris in group A
  Arms: Closed Reduction and Plaster of Paris Cast Application
Procedure: closed reduction and Percutaneous K-wire fixation and plaster of application is applied in group B — Group A Participant treated with the closed reduction and manipulation and plaster of paris application is applied for colles fracture.
  Arms: Closed Reduction with Percutaneous K-Wire Fixation and Plaster of Paris Cast Application

SUMMARY:
Colles' fracture is a common distal radius injury, often managed with closed reduction and Plaster of Paris (POP) casting. However, loss of alignment may occur with casting alone. Percutaneous K-wire fixation may improve fracture stability. This study aims to compare the functional outcomes of closed reduction with POP cast application versus closed reduction with K-wire fixation followed by POP cast application in the management of Colles' fractures.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates two commonly used treatment methods for Colles' fractures. Sixty participants were randomized into two groups: closed reduction with POP cast application, and closed reduction with percutaneous K-wire fixation followed by POP cast application. Follow-up assessments were scheduled to evaluate functional outcomes using the Gartland and Werley scoring system over a three-month period.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 60 years

Both genders

Closed Colles' fracture

Injury less than 1 week old

Provided informed consent

Exclusion Criteria:

Open fracture

Fracture with neurovascular injury

Medically unfit for surgery

Contraindication noted by orthopedic surgeon or anesthetist

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2026-01-18 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Garland and werely score | 3 months
  The Gartland and Werley scoring system (range 0-52) evaluates functional outcomes after distal radius fracture. Lower scores indicate better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Khawaja Muhammad Safdar Medical College Sialkot, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results of the primary and secondary outcomes will be shared after de-identification. Shared data will include demographic variables, baseline characteristics, and outcome measures collected during the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will be made available beginning 12 months after publication of the primary results. Data will remain available for a minimum of 5 years thereafter or until the end of the study's data-retention period, whichever occurs later
Access Criteria: Access will be granted to qualified researchers affiliated with academic, nonprofit, or governmental institutions for the purpose of scientific inquiry and secondary analyses. Researchers must submit a data-access request including a brief proposal and statistical analysis plan. Upon approval, data will be shared through a secure, controlled-access data repository. Users will be required to sign a data use agreement prohibiting re-identification or unauthorized sharing of the data
URL: https://kmsmc.edu.pk/